CLINICAL TRIAL: NCT02999256
Title: The Effect of Tart Cherry Juice Supplementation on Fat Oxidation, Body Composition and Cardio-Metabolic Markers With Cycling Exercise
Brief Title: Effect of Cherry Juice on Fat Oxidation and Cardio-metabolic Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Terun Desai, PhD Student, University of Hertfordshire
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LMS/PGT/UH/02336_
Record Dates: First submitted 2016-12-07; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Healthy; Metabolic Syndrome
Keywords: Tart Cherry Juice; Fat Oxidation; Lipid Profile; Anthocyanins; Exercise; Calorie Restrictive Mimetic
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 130ml serving twice daily (immediately before breakfast and dinner) for 20 days.
  Placebo composition: Water (100ml), Cherry Squash Concentrate (30ml), Citric Acid (1.5g), Maltodextrin (24.75g), Black Food Colouring (2ml).
  Interventions: Other: Placebo
- Montmorency Tart Cherry Juice (Experimental): 130ml serving twice daily (immediately before breakfast and dinner) for 20 days.
  MTCJ Composition: 100ml water and 30ml Montmorency tart cherry concentrate (Cherry Active, Sunbury, UK).
  Interventions: Dietary Supplement: Montmorency Tart Cherry Juice

INTERVENTIONS:
Dietary Supplement: Montmorency Tart Cherry Juice
  Arms: Montmorency Tart Cherry Juice
Other: Placebo
  Arms: Placebo

SUMMARY:
The present study examined the effect of Montmorency tart cherry juice and FATMAX (intensity eliciting maximal fat oxidation) exercise on fat oxidation rates, body composition and blood-based cardio-metabolic markers. Participants received both Montmorency tart cherry juice and placebo in a random counterbalanced order for 20 days. Outcome variables were measured immediately pre- and post-supplementation and 10 days after the onset of supplementation. It was hypothesised that Montmorency tart cherry juice would increase fat oxidation during exercise, reduce body fat percentage and improve cardio-metabolic markers.

DETAILED DESCRIPTION:
Aims: (1) Examine whether tart cherry juice supplementation with cycling exercise augments fat oxidation rate and therefore plays a role in weight management in healthy active human participants. (2) To extrapolate findings from this study to future biomedical health and disease research.

Methods: Random counterbalanced, within-group, double-blind study design. Participants were randomly allocated into consuming either cherry juice first or placebo. Eleven recreationally active male and female participants were recruited. Participants consumed 30ml Montmorency tart cherry juice concentrate mixed with 100ml water, twice daily for 20 days. Participants underwent a 14 day washout period between trials. All participants were instructed to keep to their habitual intake of polyphenols and anthocyanins. Twenty-four hours before each exercise testing session, participants consumed similar meals at the same times. Diet adherence was monitored through food diaries.

Participants attended each testing session following an overnight fast, with the testing being completed at the same time in the morning to avoid circadian variation. Preliminary testing was conducted to ascertain VO2max and individual FATMAX, 4 days before the one hour pre-supplementation exercise test. VO2max was re-assessed 4 days before the one hour post-supplementation exercise test to determine if any changes in training status affected results.

Testing will occur at baseline, 10 days after the onset of supplementation and after 20 days supplementation. Exercise protocol consisted of 60min cycling at pre-determined individual FATMAX. Continuous gas analysis and heart rate were monitored throughout. Substrate oxidation rates and energy expenditure were calculated using stoichiometric equations (Jeukendrup and Wallis, 2005). During each testing session blood pressure and body composition (impedance) measurements were taken at baseline and pre-exercise during all testing sessions. Resting metabolic rate (indirect calorimetry) was assessed at baseline and pre-exercise during all testing sessions.

Serum blood samples were obtained from participants at the following time points: baseline, pre-exercise and post-exercise for one hour submaximal exercise tests, in both trials. The following markers were analysed: Glucose, Lactate, Triglycerides, HDL, Total Cholesterol and Total Antioxidant Status.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45
* Male and Female
* Non-smokers
* Recreationally active (minimum 150 minutes physical activity per week)
* Injury free at all times of testing.

Exclusion Criteria:

* Aged <18 years old, >45 years old
* Current or previous history of gastrointestinal, cardiovascular or renal disease
* Current or previous history of injury that may be exacerbated with the exercise protocol used
* Allergy to maltodextrin or specific fruit products (especially cherries) and those currently taking medication (such as steroids, NSAIDs, antibiotics) or currently using any nutritional supplement.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Fat Oxidation (grams/min) | Pre-, Mid- (10 days) and Post- (21 days) after onset of Supplementation in both Arms

SECONDARY OUTCOMES:
Change in Lipid Profile (Total Cholesterol, HDL, Triglycerides, LDL) (mmol/L) | Pre-, Mid- (10 days) and Post- (21 days) after onset of Supplementation in both Arms
Change in Serum Glucose (mmol/L) | Pre-, Mid- (10 days) and Post- (21 days) after onset of Supplementation in both Arms
Change in Body Fat Percentage (%) | Pre-, Mid- (10 days) and Post- (21 days) after onset of Supplementation in both Arms
Change in Body Mass (kg) | Pre-, Mid- (10 days) and Post- (21 days) after onset of Supplementation in both Arms
Change in Fat Mass (kg) | Pre-, Mid- (10 days) and Post- (21 days) after onset of Supplementation in both Arms
Change in Fat Free Mass (kg) | Pre-, Mid- (10 days) and Post- (21 days) after onset of Supplementation in both Arms
Change in Total Antioxidant Status (mmol/L) | Pre-, Mid- (10 days) and Post- (21 days) after onset of Supplementation in both Arms